CLINICAL TRIAL: NCT06994377
Title: The Impact of Emotional Distress on First Line Therapy in Patients With Metastatic Breast Cancer (EIRENE): a Prospective Observational Study
Brief Title: Emotional Distress in Patients With Metastatic Breast Cancer in First Line of Therapy
Acronym: EIRENE
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: L2 - 311; UID 4907 (Other: Clinical Trial Office - Istituto Europeo di oncologia)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Emotional Distress; First Line Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A (HR-/HER2-, PD-L1+): Triple-negative Programmed Cell Death Ligand 1 (PD-L1)+ mBC patients receiving chemotherapy with immune checkpoint inhibitors (ICIs)
  Interventions: Behavioral: ED and quality of life assessment
- Cohort B (HR-/HER2-, PD-L1-): Triple-negative PD-L1- mBC patients receiving chemotherapy
  Interventions: Behavioral: ED and quality of life assessment
- Cohort C (HR+/HER2-): HR+/HER2- mBC patients receiving Cyclin-Dependent Kinase 4/6 (CDK4/6) inhibitor + endocrine therapy
  Interventions: Behavioral: ED and quality of life assessment
- Cohort D (HER2+): HER2+ mBC patients receiving chemotherapy + trastuzumab and pertuzumab
  Interventions: Behavioral: ED and quality of life assessment

INTERVENTIONS:
Behavioral: ED and quality of life assessment — Patients will undergo ED and quality of life assessments through specific questionnaires completion

SUMMARY:
Few data about the impact of emotional distress (ED) on treatment efficacy in patients with metastatic breast cancer (mBC) are available.

Aim of this study is to assess the outcomes of patients with mBC receiving first-line treatment according to the presence of baseline ED.

DETAILED DESCRIPTION:
Metastatic breast cancer (mBC) is the most incident and prevalent cancer in the world and, according to a recent meta-analysis, 50% of patients with BC report emotional distress (ED).

In patients with cancer, ED negatively impacts treatment adherence, ability to self-manage the physical and emotional consequences of cancer symptoms and treatment-related adverse events, and overall quality of life. ED has been shown to directly affect treatment outcomes in patients with breast cancer, with studies demonstrating that psychological well-being plays a critical role in therapeutic success.

Furthermore, recent studies showed that baseline ED is associated with a lower efficacy of immunotherapy in patients with non-small cell lung cancer (NSCLC) or melanoma.

Few data about the impact of ED on treatment efficacy in patients with mBC are available. In the first line setting patients receive endocrine therapy, chemotherapy, immunotherapy and/or targeted therapy according to the disease subtype. These agents display different mechanisms of action, which involve the immune system at different levels. However, the role of ED on the efficacy of these treatments according to the BC subtype is unknown.

Aim of this study is to assess the outcomes of patients with mBC receiving first-line treatment according to the presence of baseline ED.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Confirmed histological diagnosis of breast cancer
* No prior treatment for advanced/metastatic cancer
* Indication to receive first-line therapy as per standard clinical practice based on the disease subtype:

  1. cohort A (HR-/HER2-, PD-L1+): pembrolizumab or atezolizumab + chemotherapy
  2. cohort B (HR-/HER2-, PD-L1-): chemotherapy
  3. cohort C (HR+/HER2-): CDK4/6 inhibitor + endocrine therapy
  4. cohort D (HER2+): chemotherapy + trastuzumab and pertuzumab
* Presence of measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 and/or Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) criteria
* Able to provide full informed consent for the study

Exclusion Criteria:

* Pre-existing severe psychiatric disorders or other conditions that could impair the ability to provide informed consent
* Inability to complete questionnaires
* Presence of another malignancy in the previous 3 years
* Symptomatic brain metastases
* Ongoing treatment with antidepressant and/or anxiolytic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mBC eligible for standard 1st line treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS), according to the presence of ED at T0, in cohort A | 2 years
  Time from T0 (Cycle 1 Day 1) to disease progression or death

SECONDARY OUTCOMES:
Progression-free survival (PFS), according to the presence of ED at T0, in cohort B, C and D | 2 years
  Time from T0 (Cycle 1 Day 1) to disease progression or death
Progression-free survival (PFS), according to the presence of ED at T1 (Cycle 3 Day 1) | 2 years
  Time from T0 (Cycle 1 Day 1) to disease progression or death
Objective response rate (ORR), according to the presence of ED at T0 and T1 | 2 years
  Number of partial response or complete response achieved
Quality of life evaluation | 3 months
  Completion of European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) EORTC-QLQ-C30 (minimum value: 1, maximum value: 4 - higher scores mean a greater agreement with the statement)
Fear of cancer progression evaluation | 3 months
  Completion of Fear of Progression Questionnaire (FoP Q) (minimum value: 1, maximum value: 5 - higher total score reflects a higher level of fear of disease progression)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, MD, PhD, Principal Investigator — European Istitute of Oncology
Locations (36):
- Italy (36):
  - Ospedali Riuniti di Ancona, Ancona
  - CRO (Centro di Riferimento Oncologico), Aviano
  - Azienda Usl Toscana centro - Ospedale Santa Maria Annunziata, Bagno a Ripoli
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - ASST Spedali Civili, Brescia
  - Ospedale A. Perrino, Brindisi
  - ASST della Valle Olona, Busto Arsizio
  - Ospedale Valduce, Como
  - Ospedale Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - AOU Gaetano Martino di Messina, Messina
  - European Institute of Oncology, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale Niguarda, Milan
  - Ospedale San Giuseppe MultiMedica, Milan
  - Policlinico di Milano, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Ospedale Maggiore di Novara, Novara
  - Policlinico Universitario Paolo Giaccone, Palermo
  - Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Usl Toscana centro - Ospedale di Prato Santo Stefano, Prato
  - Ospedale Infermi, Rimini
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Policlinico Umberto I, Rome
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
  - ASL CN2 - Ospedale Michele e Pietro Ferrero, Verduno
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
  - Ospedale Sacro Cuore Don Calabria - Negrar, Verona
  - ASST Brianza, Vimercate